CLINICAL TRIAL: NCT04825327
Title: Predicting the Future: Incipient Tuberculosis
Acronym: PreFIT
Status: Completed | Type: Observational
Sponsor: Amsterdam Institute for Global Health and Development (Other)
Collaborators: University of Stellenbosch (Other); Makerere University (Other); Centro de Investigacao em Saude de Manhica (Other); Barcelona Institute for Global Health (Other); Foundation for Innovative New Diagnostics, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: RIA2018D-2509
Record Dates: First submitted 2021-03-28; First posted 2021-04-01 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Tuberculosis
Keywords: Diagnostic accuracy; Host response cartridge; TB contacts; Incipient TB; Point-of-care-testing
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Fingerprick blood for point-of-care testing, two serum tubes, one Tempus RNA tube, urine (30ml) and sputum (max 3 sputa) will be collected from cohort participants who are TB presumptive or meeting sputum expectorator definition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators will study, prospectively, if contacts (household or close contacts) of tuberculosis (TB) patients with high C-reactive protein (CRP), low hemoglobin (Hb) levels, and a positive Xpert Host Response (HR) cartridge result develop active TB within 12 months. They will also investigate if there is a correlation between progressing to active TB within 12 months and having high levels of the iron homeostasis markers (Hepcidin, Ferritin and Transferrin).

Identified index cases who agree to participate will refer their household or close contacts to also join the study. These contacts will be tested for TB and only contacts who are negative will be enrolled and followed-up at 6 months and 12 months. Blood samples will be collected at baseline and 6 months for testing. During the study period, TB testing will be done on contacts who meet symptoms criteria. At 12 months, all contacts will undergo a chest x-ray to assist in the diagnosis of TB.

PreFIT will target people aged 12 to 60 years of age and both HIV negative and positive. 1515 trial participants will be recruited at Stellenbosch University in South Africa, 1515 at Fundaçao Manhiça in Mozambique and 1010 at Makerere University in Uganda, respectively.

DETAILED DESCRIPTION:
Although the estimated numbers of people infected with TB in Africa are declining since the rollout of antiretroviral therapy a decade ago, TB is still the highest in the world. Early diagnosis and treatment of TB disease are essential to reducing morbidity and mortality. Transformative progress will never be possible with the current diagnostic tools as they rely on the detection of active TB which usually happen after disease has already been spread to others. Diagnostic technologies to accurately detect who will develop active TB are under development. However, their performance is not well reported.

A better TB prediction test is needed to detect TB before clinical manifestation. The PreFIT investigators hypothesize that volunteers with a combination of positive Xpert HR result, high CRP, and/or low Hb levels will likely progress to active TB within 12 months. They also hypothesize that those with TB will have early high Hepcidin, Ferritin and Transferrin levels.

The investigators plan to ask those found with TB at the local clinic if they accept to join the study. The participants, if they consent will then give information about people (contacts) who they stay with or meet frequently to also join the study. Contacts who have TB symptoms will be asked to cough sputum to be tested for co-prevalent TB disease. If they are found not to have TB disease, they will be asked to give blood: few drops from a finger prick and about 50mls from the vein on the arm to be stored and used for further tests. Follow-up and sampling of enrolled contacts without co-prevalent active TB will occur at six and 12 months (± 21 days before or after each time point, a six-week total window). Participants meeting presumptive TB or sputum expectorator definitions at six (M6) or 12 months (M12) of follow-up, or report with symptoms at any timepoint in-between, will undergo Xpert Ultra (or Xpert MTB/RIF if Ultra unavailable) and culture testing. All positive cultures will undergo whole genome sequencing (WGS) to track index case and co-prevalent or incident case transmission. Chest X-ray (CXR) will be done at M12 to potentially rule-out active disease missed by microbiological methods. Passive TB diagnoses (microbiological or empirical) throughout the follow-up period will be captured.

To prevent diagnostic information bias, M0 and M6 test results for Xpert HR, CRP and haemoglobin will be kept concealed to the study nurse(s) and physician(s) who screen the cohort participants for active TB during follow-up. Similarly, laboratory technicians who test the stored samples for hepcidin, transferrin and ferritin will be blinded to whether the sample is from a participant who developed active TB during follow-up, or from a cohort participant who did not.

The study will recruit 1515 trial participants each at Stellenbosch University in South Africa, 1515 at Centro de Investigação em Saúde de Manhiça in Mozambique and 1010 at Makerere University in Uganda. Participants will be between the ages of 12 and 60 years; pregnant women, minorities, economic and education disadvantaged, both HIV negative and positive will join the study. Contacts found to have co-prevalent active TB, potential pathologies on CXR, abnormal Hb and CRP levels will be referred to the local clinic for investigation per standard-of-care with a written summary of the relevant study results. All participant information will be treated in a strictly confidential manner and will be identified only by a code and not by any personal identifier.

PreFIT's results will contribute to the development and uptake of accurate, cost-effective, scalable and field-friendly diagnostic tools, to facilitate scale-up of preventive treatment in sub-Saharan Africa and beyond.

ELIGIBILITY:
Inclusion Criteria:

Index cases

1. ≥18 years old
2. Willing to provide the contact information of people who meet the definition of contacts, or willing to refer those people (which make require the distribution of study pamphlets) so that may contact study staff
3. Willing to comply with study requirements i.e. provision of contact details and written, informed consent prior to enrolment
4. Willing to provide sputa (expectorated or induced) for culture; and
5. Meeting the definition for active TB.

Contacts (cohort)

1. ≥12 years old
2. Meeting contact definition
3. Able and willing to return for follow-up visits, with no plans to move soon
4. Willing to comply with study requirements i.e. provision of contact details and written, informed consent or assent prior to enrolment
5. Willing and able to provide sputum and blood
6. Agree to potentially undergo CXR at M12 (women

Exclusion Criteria:

Index cases

1. No informed consent or assent
2. More than six weeks has passed since the index case's first bacteriological result for TB was reported
3. Patient was started on treatment based on empirical or clinical grounds (including CXR) alone
4. Patient with rifampicin resistance (known from Xpert, Ultra, and/or MTBDRplus results)

Contacts (cohort)

1. No informed consent or assent
2. Not diagnosed with active TB
3. Unwilling or unable to provide blood
4. More than six weeks has passed since reporting of the index case's first positive test result
5. Has taken any form of TB treatment within the preceding two months (i.e., is currently on treatment). There are no exclusions based on any TB treatment more than two months prior.

Ages: 12 Years to 60 Years | Sex: All
Age Groups: Child, Adult
Study Population: Presumptive TB patients diagnosed by the TB programme or as part of an ongoing study with bacteriologically confirmed (smear microscopy, Xpert, Ultra, culture, or MTBDRplus) active TB, and any person who has been exposed to the presumptive TB patients will be recruited from primary care clinics.
  The presumptive TB patients are enrolled to find and select the exposed individuals who will constitute the cohort.
Sampling Method: Non-Probability Sample
Enrollment: 3016 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Predictive accuracy of each assay for incident TB occurring over a 12-month period from enrolment. | 12 months
  Predictive accuracy is operationalized in the following metrics: sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV), for each assay at a predefined cut-off value for a positive versus negative test result.

SECONDARY OUTCOMES:
Assay turnaround time and error rates | 30 months
  Point-of-care or near-point-care feasibility for the prospectively validated assays
Accuracy of predictive algorithms | 12 months
  Sensitivity, specificity, PPVs, and NPVs of different combinations of tests, done concurrently or sequentially ("diagnostic algorithms")
Diagnostic cost | 12 months
  Total diagnostic cost per incident case of active TB correctly predicted using an established bottom-up micro-costing methodology developed and validated for TB

CONTACTS AND LOCATIONS:
Overall Officials: Grant Theron, PhD, Principal Investigator — University of Stellenbosch; Alberto L Garcia-Basteiro, PhD, Study Director — Barcelona Institute for Global Health; Adam Penn-Nicholson, PhD, Study Director — The Foundation for Innovative New Diagnostics
Locations (3):
- Centro de Invesigação em Saúde de Manhiça, Manhiça, Mozambique
- University of Stellenbosch, Cape Town, South Africa
- Makerere University, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Collaborators will have access to de-identified IPD data. Other researchers wishing to access the data will be required to sign a data sharing agreement as per institutional policies.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be available once the findings are published.
Access Criteria: Data access will be granted to interested collaborators and parties through sharing of data files or login information for the study's secure RedCap electronic database during the course of patient recruitment.

REFERENCES:
- See also: project website — http://predictingtb.org/